CLINICAL TRIAL: NCT04451135
Title: Correlating Electroconvulsive Therapy Response to Electroencephalographic Ictal Complexes and Postictal Markers
Brief Title: CET- REM (Correlating ECT Response to EEG Markers)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202006108
Record Dates: First submitted 2020-06-24; First posted 2020-06-30 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: ECT; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Treatment-Resistant Depression (Experimental)
  Interventions: Diagnostic Test: Electroencephalographic (EEG); Diagnostic Test: Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR16); Diagnostic Test: Ictal Electroencephalographic (EEG) Measurements; Diagnostic Test: Post-Ictal Electroencephalographic (EEG) Suppression Measurements

INTERVENTIONS:
Diagnostic Test: Electroencephalographic (EEG) — EEG on nights after ECT session will be recorded using the DREEM device. Sleep EEG data will also be acquired for a minimum of one night prior to the first ECT session, providing a true baseline measure. The DREEM device allows continuous recording of multichannel EEG
Diagnostic Test: Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR16) — The Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR16) is a measure of depression symptom severity that has been validated for clinical and research use53. It is a standard self-report measurement completed by patients prior to each ECT session
Diagnostic Test: Ictal Electroencephalographic (EEG) Measurements — A high-density 65-electrode EEG scalp electrode net (EGI/Philips) with Elefix conductive gel injected within Ag/AgCl electrode sensors is utilized to monitor brain activity during the ictal period
Diagnostic Test: Post-Ictal Electroencephalographic (EEG) Suppression Measurements — A board-certified epileptologist will review all seizures to assess seizure parameters, including duration of seizure and interval of PGES. Preprocessing of the PGES periods will be accomplished with band-pass filtering from 2 to 30 Hz with 1st order Butterworth filters.

SUMMARY:
Single-center study to determine the relationship between changes in depression symptoms and electroencephalographic (EEG) patterns induced by electroconvulsive therapy (ECT)

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) is an effective treatment for many psychiatric illnesses, including major depressive disorder. While effective, objective markers have not been developed to predict clinical outcome trajectories following ECT. This is important given the risks and costs incurred during a full treatment course. Electroencephalography (EEG) is typically employed to monitor the generation and termination of ECT-induced seizures but leverage of markers toward prognostication remains a future goal. The investigators have characterized two distinct EEG patterns associated with ECT-induced generalized seizures and have two sleep markers that may serve as markers for predicting response to treatment. Central Positive Complexes (CPCs) are large ictal complexes with a scalp topology of voltage declining from the top of the head. CPCs are localized to cortical areas that are involved in the formation of sleep spindles and slow wave sleep. A pattern of low-voltage activity, known as post-ictal generalized electroencephalographic suppression (PGES), is frequently used to document termination of these seizures. Additionally, two EEG markers of sleep microstructure may have utility given their association with synaptic plasticity, a process presumably invoked over the course of ECT-induced recovery from psychiatric illness as pathologic neural circuitry undergoes reconfiguration. These two markers, sleep spindles and slow waves show altered expression patterns in patients with psychiatric disorders, and thus may be useful as objective markers of ECT responsiveness. None of the above EEG markers have been explored for an association to interval changes in disease severity over the course of ECT. This project will incisively probe the relationships between temporal trajectories of major depressive disorder severity and longitudinal measurements of ictal and postictal EEG markers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Referral for ECT index course for treatment-resistant depression (unipolar major depressive disorder or bipolar depression), major depressive disorder with psychotic symptoms, schizophrenia or schizoaffective being treated for a depressed episode, unspecified depression

Exclusion Criteria:

* Schizophrenia or schizoaffective disorder not being treated for a depressed episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Interval change in Quick Inventory of Depressive Symptomatology-16 Item Self Report (QIDS-SR16) between ECT sessions. | Up to 8 weeks during patients ECT treatment course
  16 item Self-report questionnaire that best describes the participant's depressive symptoms over the last seven days. Scale: 0=never or do not, 3=nearly all the time, or the highest level of time listed on the question.
Duration of Central Positive Complexes during ECT treatments. | Up to 8 weeks during patients ECT treatment course
  Total time (in seconds) during the ictal period for which CPCs are present in the EEG immediately following seizure induction until termination of the seizure.
  Range of values: 0 - 300 seconds
Duration of PGES during ECT treatments. | Up to 8 weeks during patients ECT treatment course
  Total time (in seconds) during the postictal period for which PGES is present in the EEG immediately following seizure termination for up to 5 minutes.
  Range of values: 0 - 300 seconds
Density of EEG sleep spindles during non-rapid eye movement (NREM) stages N2 on evenings following ECT treatments. | Up to 8 weeks during patients ECT treatment course
  The total number of EEG sleep spindles per minute present during N2 sleep. Range of values: 0 - 60 spindles/min
Slow wave activity (SWA) during N3 sleep on evenings following ECT treatments | Up to 8 weeks during patients ECT treatment course
  Total power of EEG slow waves per minute present during the first identified cycle of N3 sleep Range of values: 0 - 50 dB/min

CONTACTS AND LOCATIONS:
Overall Officials: MohammadMehdi Kafashan, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Lopez J, Hoffmann R, Armitage R. Reduced sleep spindle activity in early-onset and elevated risk for depression. J Am Acad Child Adolesc Psychiatry. 2010 Sep;49(9):934-43. doi: 10.1016/j.jaac.2010.05.014. Epub 2010 Jul 24. PMID 20732629
- [Background] Kho KH, van Vreeswijk MF, Simpson S, Zwinderman AH. A meta-analysis of electroconvulsive therapy efficacy in depression. J ECT. 2003 Sep;19(3):139-47. doi: 10.1097/00124509-200309000-00005. PMID 12972983
- [Derived] Kafashan M, Brian Hickman L, Labonte AK, Huels ER, Maybrier H, Guay CS, Subramanian S, Farber NB, Ching S, Hogan RE, Kelz MB, Avidan MS, Mashour GA, Palanca BJA. Quiescence during burst suppression and postictal generalized EEG suppression are distinct patterns of activity. Clin Neurophysiol. 2022 Oct;142:125-132. doi: 10.1016/j.clinph.2022.07.493. Epub 2022 Jul 30. PMID 36030576